CLINICAL TRIAL: NCT02304042
Title: Carbetocin Versus Oxytocin in the Prevention of Post Partum Haemorrhage (PPH) in Women Delivered Vaginally With at Least 2 Risk Factors for Atonic PPH: A Randomised Controlled Trial
Acronym: PPH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PPH 2
Record Dates: First submitted 2014-11-26; First posted 2014-12-01 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Delivery
MeSH Terms: interventions — carbetocin; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carbetocin (Active Comparator): 125 women will receive carbetocin after delivery of the anterior shoulder. The drug will be diluted in 10ml saline and will be given by the slowly intravenously after delivery of the anterior shoulder
  Interventions: Drug: Carbetocin
- Oxytocin (Active Comparator): 125 women will receive carbetocin oxytocin after delivery of the anterior shoulder. The drug will be diluted in 10ml saline and will be given by the slowly intravenously after delivery of the anterior shoulder
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Carbetocin — Carbetocin will be given slowly iv after delivery of the anterior shoulder.
  Arms: Carbetocin
Drug: Oxytocin — Oxytocin will be given slowly iv after delivery of the anterior shoulder.
  Arms: Oxytocin

SUMMARY:
250 women will be randomly divided into 2 equal groups using computer generated random numbers. Group 1 will receive Carbetocin 100 µgm (Pabal® Ferring, UK) and group 2 will receive oxytocin 5IU (Syntocinon®, Novartis, Switzerland). Both drugs will be diluted in 10ml saline and will be given by the slowly intravenously after delivery of the anterior shoulder. The investigators will not include a control group for ethical reasons.

DETAILED DESCRIPTION:
Obstetric haemorrhage remains one of the major causes of maternal death in both developed and developing countries (1). Postpartum haemorrhage (PPH) is defined as a blood loss >500 ml more of blood from the genital tract within 24 hours of the birth of a baby. PPH can be minor (500-1000 ml) or major (more than 1000 ml). The most frequent cause of PPH is uterine atony, contributing up to 80 % of the PPH cases.

Risk factors of atonic PPH include multiple pregnancy, placenta previa, previous PPH, body mass index (BMI) >30, prolonged labour, fetal macrosomia>4kg and primipara> 40 years.

Oxytocin is currently the uterotonic of first choice. It has proven to decrease the incidence of PPH by 40 % and has a rapid onset of action and a good safety profile. A disadvantage of oxytocin is its short half-life of 4-10 min, regularly requiring a continuous intravenous infusion or repeated intramuscular injections.

Carbetocin is a long-acting oxytocin analogue indicated for the prevention of uterine atony after child birth by CS under epidural or spinal anaesthesia. Carbetocin has a rapid onset of action (within 1-2 min) and a prolonged duration of action (approximately 1 h) because of sustained uterine response with contractions of higher amplitude and frequency. Its safety profile is comparable to that of oxytocin.

The study will be conducted in Cairo university hospitals and BeniSuef university hospitals. All patients with at least 2 risk factors for developing atonic PPH will be approached in the antenatal clinic or early in labour if appropriate. Risk factors include previous PPH, BMI>35, multiple pregnancy, prolonged labour >12 hours, fetal macrosomia>4kg and induction of labour. Women will be invited to participate in the study, the invitation will include a clear full explanation of the study. Only patients signing informed written consents will participate in the study.

250 women will be randomly divided into 2 equal groups using computer generated random numbers. Group 1 will receive Carbetocin 100 µgm (Pabal® Ferring, UK) and group 2 will receive oxytocin 5IU (Syntocinon®, Novartis, Switzerland). Both drugs will be diluted in 10ml saline and will be given by the slowly intravenously after delivery of the anterior shoulder. We will not include a control group for ethical reasons.

The uterine tone and amount of bleeding will be noted and the need for further uterotonic agents will be determined 2 minutes after giving the drug. Blood loss will be estimated through weighing the swabs and using pictorial charts. Blood haemoglobin will be assessed 24 hours after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women with at least 2 risk factors for developing PPH. Risk factors include previous PPH, BMI>35, multiple pregnancy, prolonged labour >12 hours, ultrasound estimated fetal weight>4kg and induction of labour.

Exclusion Criteria:

* Gestational age <37 weeks
* Placenta previa
* Hypertension.
* Preeclampsia.
* Cardiac, renal or liver diseases
* Known hypersensitivity to Carbetocin.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Need for other uterotonics | 2 minutes after giving the drug
  After giving the drug, the uterine tone will be felt and amount of bleeding will be estimated.

SECONDARY OUTCOMES:
Bleeding>500ml | 2 minutes after giving the drug.
  The amount of bleeding will be estimated 2 minutes after giving the drug.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - BeniSuef University hospitals, BeniSuef
  - Cairo University Hospitals, Cairo

REFERENCES:
- [Background] Winter C, Macfarlane A, Deneux-Tharaux C, Zhang WH, Alexander S, Brocklehurst P, Bouvier-Colle MH, Prendiville W, Cararach V, van Roosmalen J, Berbik I, Klein M, Ayres-de-Campos D, Erkkola R, Chiechi LM, Langhoff-Roos J, Stray-Pedersen B, Troeger C. Variations in policies for management of the third stage of labour and the immediate management of postpartum haemorrhage in Europe. BJOG. 2007 Jul;114(7):845-54. doi: 10.1111/j.1471-0528.2007.01377.x. PMID 17567419
- [Background] Moertl MG, Friedrich S, Kraschl J, Wadsack C, Lang U, Schlembach D. Haemodynamic effects of carbetocin and oxytocin given as intravenous bolus on women undergoing caesarean delivery: a randomised trial. BJOG. 2011 Oct;118(11):1349-56. doi: 10.1111/j.1471-0528.2011.03022.x. Epub 2011 Jun 14. PMID 21668768